CLINICAL TRIAL: NCT04979585
Title: Camrelizumab Combined With Anlotinib and Nab-paclitaxel in Patients With Untreated Advanced Mucosal Melanoma:a Single-arm, Multicenter, Open-label Study
Brief Title: Camrelizumab Plus Amlotinib and Chemotherapy in the First-line Treatment of Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Di Wu (Other)
Responsible Party: Sponsor-Investigator, Di Wu, Professor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-ME-01
Record Dates: First submitted 2021-04-26; First posted 2021-07-28 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — camrelizumab; anlotinib; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: camrelizumab combined with anlotinib and nab-paclitaxel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients with untreated advanced mucosal melanoma
  Interventions: Drug: Camrelizumab; Drug: Anlotinib; Drug: nab-Paclitaxel

INTERVENTIONS:
Drug: Camrelizumab — 200mg ,IV,d1,Q3W.
Drug: Anlotinib — 8mg,oral, d1-14,Q3W.
Drug: nab-Paclitaxel — 260mg/m2,IV,d1,Q3W.

SUMMARY:
To evaluate the objective response rate of camrelizumab combined with anlotinib and nab-paclitaxel in patients with untreated advanced mucosal melanoma.

DETAILED DESCRIPTION:
The current traditional cytotoxic single agent or combination chemotherapy cannot clearly improve the overall survival rate of patients with advanced melanoma.From the current point of view, combination therapy will be one of the inevitable trends in the future development of tumor immunotherapy. So carry out this research To evaluate the objective response rate of camrelizumab combined with anlotinib hydrochloride and albumin paclitaxel in the first-line treatment of patients with advanced mucosal melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender ;
2. It was confirmed by histopathology that patients with recurrence, unresectable or metastatic mucosal melanoma after surgery (stage III/IV).
3. Have not received any systemic anti-tumor drug therapy in the past, and allow previous adjuvant therapy or neoadjuvant therapy (except PD-1/PDL1 monoclonal antibody and VEGFR TKI), but it is required to be completed at least 4 weeks before the first administration of the study drug, and All related toxic events have returned to normal or CTCAE4.03 grade I or below, except for hair loss).
4. ECOG 0or1。
5. The expected survival time is ≥12 weeks.
6. Can swallow medicine normally.
7. According to the RECIST 1.1 standard, there is at least one measurable lesion, and the lesion has not been irradiated.
8. Patients are allowed to have a history of brain/meningeal metastasis, but they must undergo local treatment (surgery/radiotherapy) before the start of the study, and be clinically stable for at least 3 months (allowing corticosteroids before the first use of the study drug, but before starting the study drug Need to stop for 2 weeks);
9. Patients have good organ function: no blood transfusion or collection stimulation factors and plateplate production in the 14 days before the first drug was given, neutral granulocyte count ≥1.5×109/L, plate count≥ × 80×109/L, hemoglobin ≥80 g/L, serum creatinine ≤1.5x normal upper limit (ULN), total bilium ≤1.5x normal upper limit Value (ULN) ALT, AST≤2.5x ULN (no liver transfer) or ≤5x ULN (e.g. liver transfer), albumin ≥30 g/L, blood clotting function requirements: international standardized ratio Value (INR≤ 1.5x ULN, coagulase original time (PT) ≤1.5x ULN, active partial clotting enzyme time (APTT) ≤1.5x ULN. Electrolyte requirements: corrected serum calcium, blood potassium,
10. Women of childbearing age must have a negative serum pregnancy test result within 7 days before the first administration of the trial drug; reproductive men or women who are likely to become pregnant must use highly effective contraceptive methods (such as oral contraceptives, uterine contraceptives, etc.) during the entire trial. Internal contraceptive device, sexual desire control or barrier contraception combined with spermicide), and continue contraception for 12 months after the end of treatment.
11. The subjects voluntarily joined the study, signed an informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. Patients who have previously received anti-PD-1, anti-PD-L1, anti-PD-L2 therapy and or VEGFR TKI therapy.
2. Patients currently undergoing anti-tumor therapy.
3. Patients who have participated in or are participating in clinical trials of other drugs/therapies within 4 weeks before the first use of the study drug.
4. The study drug has undergone a major surgical operation or has not recovered from the side effects of this operation within 4 weeks before the first administration of the study drug, live vaccination, immunotherapy, and radiotherapy within 2 weeks
5. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, thyroid Hyperfunction; patients suffering from vitiligo; asthma has been completely relieved in childhood, and can be included in adults without any intervention; patients with asthma that require bronchodilators for medical intervention cannot be included).
6. The patient is using immunosuppressive agents or systemic hormone therapy to achieve immunosuppressive purposes (dose>10mg/day prednisone or other curative hormones), and continues to use it within 2 weeks before enrollment.
7. In the past 5 years, there is a history of other malignant tumors other than mucosal melanoma, except for cured skin basal cell carcinoma, skin squamous cell carcinoma, early prostate cancer and cervical carcinoma in situ.
8. Patients who have received hematopoietic stimulating factors, such as granulocyte colony stimulating factor (G-CSF), erythropoietin, etc., within 1 week before the first administration of the study drug.
9. The HIV antibody or Treponema pallidum antibody test result is positive.
10. Patients with active hepatitis B or C: If HBsAg or HBcAb is positive, add HBV DNA (the test result is higher than the upper limit of the normal range). If the HCV antibody test result is positive, add HCV RNA (the test result is higher than the upper limit of the normal range).
11. Those who are known to be allergic to recombinant humanized PD-1 monoclonal antibody drugs and their components; those who are known to be allergic to anlotinib and any of its excipients; those who are known to be allergic to albumin paclitaxel and its excipients.
12. A large amount of pleural fluid or ascites with clinical symptoms that require symptomatic treatment.
13. Active lung disease (interstitial pneumonia, pneumonia, obstructive lung disease, asthma) or a history of active tuberculosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-04-14 (Estimated); Study Completion 2023-08-14 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  defined as the proportion of patients whose tumor volume has shrunk to a predetermined value and can maintain the minimum time limit. The sum of complete remission plus partial remission.

SECONDARY OUTCOMES:
PFS | 1 year
  The time from the beginning of randomization to the onset of disease progression or the death of the patient.

OTHER OUTCOMES:
DCR | 1 year
  The percentage of cases that achieved remission (PR+CR) and stable disease (SD) after treatment accounted for the number of evaluable cases.

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No